CLINICAL TRIAL: NCT03291288
Title: An Open-label, Single Sequence, Crossover Drug-drug Interaction Study Assessing the Effect of Pexidartinib on the Pharmacokinetics of CYP3A4 and CYP2C9 Substrates in Patients
Brief Title: Effect of Pexidartinib on the Way the Body Processes CYP3A4 and CYP2C9 Substrates (Pharmacokinetics)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PL3397-A-U126
Record Dates: First submitted 2017-09-19; First posted 2017-09-25 (Actual); Results first posted 2020-03-19 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-04

CONDITIONS: Drug Interaction Potential
Keywords: Tenosynovial Giant Cell Tumors (TGCT); Kit-mutant melanoma; Kit-mutant gastrointestinal stromal tumor (GIST); Cocktail drug-drug interaction (DDI)
MeSH Terms: conditions — Synovitis, Pigmented Villonodular | interventions — Tolbutamide; Midazolam; Bro protein, Drosophila; pexidartinib

STUDY DESIGN:
Intervention Model Description: Open-label, single sequence study with 2 parts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pexidartinib (Experimental): Part 1 (Drug-drug Interaction Phase):
  On Day 1, all participants will receive a single oral dose each of midazolam (2 mg) and tolbutamide (500 mg). On Day 3, pexidartinib (800 mg/d) in twice daily (400 mg BID) dosing will be initiated and continue throughout the remainder of Part 1 and into Part 2. On the first day of pexidartinib treatment (Day 3), a single dose of midazolam (2 mg) and tolbutamide (500 mg) will be co-administered with the morning pexidartinib dose (400 mg). On Day 13, a single dose of midazolam (2 mg) and tolbutamide (500 mg) will be co-administered with the morning dose of pexidartinib (400 mg).
  Part 2 (Efficacy and Safety Phase):
  All participants will continue to receive pexidartinib 400 mg BID.
  Interventions: Drug: Tolbutamide; Drug: Midazolam; Drug: Pexidartinib

INTERVENTIONS:
Drug: Tolbutamide — Commercially available tolbutamide
  Other Names: Orinase
Drug: Midazolam — Commercially available midazolam
  Other Names: Dormicum; Hypnovel; Versed; Others
Drug: Pexidartinib — Pexidartinib is formulated as opaque, white, 200-mg capsules
  Other Names: PLX-3397

SUMMARY:
This study has two parts.

Part 1 will evaluate how pexidartinib affects the way the body processes CYP3A4 and CYP2C9 substrates using midazolam and tolbutamide, respectively, as probe agents.

Part 2 will test the efficacy and safety of pexidartinib treatment in various tumor types.

In Part 2, the same participants will continue to receive pexidartinib twice daily.

Participants will be allowed to continue using pexidartinib as long as the participant derives benefit.

ELIGIBILITY:
Inclusion Criteria:

* Is the age of majority in country of residence
* Has a diagnosis of:

  1. tenosynovial giant cell tumor (TGCT), which is associated with severe morbidity or functional limitations and for whom surgery is not an option (prior pexidartinib is permitted for TGCT patients unless ineffective or not tolerated and there has been a washout period of at least 4 weeks)
  2. KIT-mutant tumor, including melanoma or gastrointestinal stromal tumor (GIST), for which there is no standard systemic therapy, or
  3. other solid tumors (all comers) for which there is no standard systemic therapy and there is a rationale for use of pexidartinib at the Investigator's discretion
* If a female of childbearing potential, had a negative serum pregnancy test within 14 days before enrollment, or within 72 hours before enrollment where required
* Is a non-sterile male or female willing to use of one of the protocol-defined highly effective contraception methods:

  1. intra-uterine device (nonhormonal or hormonal)
  2. sexual abstinence (only if this is in line with the patient's current lifestyle)
  3. barrier methods (eg, condom, diaphragm) used in combination with hormonal methods associated with inhibition of ovulation
* Is a surgically sterile male or female, or is postmenopausal for at least 1 year, at least 50 years of age, with a follicle-stimulating hormone level > 40 milli-International units per mL (mIU/mL)
* Has adequate hematologic, hepatic, and renal function as defined by the protocol
* Is able and willing to follow all study procedures
* Has provided a signed informed consent

Exclusion Criteria:

* Is pregnant or breastfeeding
* Is unable to swallow oral medication
* Is unable to follow study procedures
* Is taking or has taken any medications or therapies outside of protocol-defined parameters
* Has any disease or condition that, per protocol or in the opinion of the investigator, might affect:

  1. safety and well-being of the participant or offspring
  2. safety of study staff
  3. analysis of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2021-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Chair — Daiichi Sankyo
Locations (11):
- United States (8):
  - HonorHealth, Scottsdale, Arizona
  - University of Arizona, Tucson, Arizona
  - Stanford University, Palo Alto, California
  - University of Kansas Cancer Center, Westwood, Kansas
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Center, Detroit, Michigan
  - Northwell Health, Lake Success, New York
  - Mary Crowley Cancer Research, Dallas, Texas
- Leids Universitair Medisch Centrum, Leiden, Netherlands
- Christchurch Hospital NZ, Christchurch, New Zealand
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Lewis JH, Gelderblom H, van de Sande M, Stacchiotti S, Healey JH, Tap WD, Wagner AJ, Pousa AL, Druta M, Lin CC, Baba HA, Choi Y, Wang Q, Shuster DE, Bauer S. Pexidartinib Long-Term Hepatic Safety Profile in Patients with Tenosynovial Giant Cell Tumors. Oncologist. 2021 May;26(5):e863-e873. doi: 10.1002/onco.13629. Epub 2020 Dec 24. PMID 33289960

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 32 participants who met all inclusion and no exclusion criteria were enrolled in the study; 2 participants did not receive pexidartinib treatment.
Pre-assignment Details: This open-label, single sequence crossover study comprised of 2 parts. Part 1 was the initial single sequence crossover part to evaluate the effect of pexidartinib on the pharmacokinetics of midazolam and tolbutamide, the drug-drug interaction (DDI) phase. Part 2 was an evaluation of efficacy and safety of pexidartinib treatment in various tumors.
Groups:
- Part 1: Drug-drug Interaction Phase: On Day 1, participants received the single oral dose of midazolam (2 mg) and tolbutamide (500 mg).
  On Day 3, pexidartinib (800 mg/day) administered as 400 mg twice daily (BID) was initiated and continued throughout the remainder of Part 1 and into Part 2. On the first day of pexidartinib treatment (Day 3), a single dose of midazolam (2 mg) and tolbutamide (500 mg) was co-administered with the morning pexidartinib dose (400 mg).
  On Day 13, a single dose of midazolam (2 mg) and tolbutamide (500 mg) was co-administered with the morning dose of pexidartinib (400 mg).
- Part 2: Pexidartinib Only: All participants received pexidartinib twice daily (BID) dosing in 28-day cycles at the 400 mg/day dose for up to one year.
Period: Drug-drug Interaction Phase
Arm/Group | Part 1: Drug-drug Interaction Phase | Part 2: Pexidartinib Only
Started | 32 | 0
Completed | 26 | 0
Not Completed | 6 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Disease progression | 1 | 0
Not completed — Other | 3 | 0
Period: Pexidartinib Only
Arm/Group | Part 1: Drug-drug Interaction Phase | Part 2: Pexidartinib Only
Started | 0 (This is a crossover trial; participants who completed Part 1 continued to Part 2.) | 26
Completed | 0 | 24
Not Completed | 0 | 2
Not completed — Ongoing | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants who received pexidartinib in Part 1 and Part 2 of the study.
Arm/Group | All Participants
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 19
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (19.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Analysis: Maximum Concentration (Cmax) for Midazolam
Description: Plasma samples for midazolam were collected at predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 24, and 48 hours (h) (±10 minutes up to 1 h, ±10% thereafter) on Days 1 to 3, and also when co-administered with pexidartinib on Days 3 (to 5) and Days 13 (to 15).
Time Frame: Baseline to 15 days post treatment
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Evaluable population.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Part 1: Midazolam Only: All participants received a single oral dose of midazolam (2 mg) on Day 1.
- Part 1: Pexidartinib + Midazolam (Cycle 1, Day 1); Part 1: Pexidartinib + Midazolam (Cycle 1, Day 11): All participants received a single oral dose of midazolam (2 mg) on Day 3 concomitantly with pexidartinib and on Day 13 following approximately 10 days of pexidartinib twice daily (BID) dosing.
Arm/Group | Part 1: Midazolam Only | Part 1: Pexidartinib + Midazolam (Cycle 1, Day 1) | Part 1: Pexidartinib + Midazolam (Cycle 1, Day 11)
Number analyzed (Participants) | 32 | 30 | 25
ng/mL | 13.6 (6.8) | 12.0 (4.9) | 9.7 (4.1)

2. Primary Outcome: Pharmacokinetic Analysis: Maximum Concentration (Cmax) for Tolbutamide
Description: Plasma samples for tolbutamide were collected at predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 24, and 48 h (±10 min up to 1 h, ±10% thereafter) on Days 1 to 3, and also when co-administered with pexidartinib on Days 3 (to 5) and Days 13 (to 15).
Time Frame: Baseline to 15 days post treatment
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Evaluable population.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Part 1: Tolbutamide Only: All participants received a single oral dose of tolbutamide (500 mg) on Day 1.
- Part 1: Pexidartinib + Tolbutamide (Cycle 1, Day 1); Part 1: Pexidartinib + Tolbutamide (Cycle 1, Day 11): All participants received a single oral dose of tolbutamide (500 mg) concomitantly with pexidartinib and on Days 3 and 13 following approximately 10 days of pexidartinib twice daily (BID) dosing.
Arm/Group | Part 1: Tolbutamide Only | Part 1: Pexidartinib + Tolbutamide (Cycle 1, Day 1) | Part 1: Pexidartinib + Tolbutamide (Cycle 1, Day 11)
Number analyzed (Participants) | 32 | 30 | 25
ng/mL | 44400 (13100) | 46700 (16300) | 44400 (12200)

3. Primary Outcome: Pharmacokinetic Analysis: Time to Maximum Concentration (Tmax) for Midazolam
Description: as for outcome 1
Time Frame: Baseline to 15 days post treatment
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Evaluable population.
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1: Midazolam Only | Part 1: Pexidartinib + Midazolam (Cycle 1, Day 1) | Part 1: Pexidartinib + Midazolam (Cycle 1, Day 11)
Number analyzed (Participants) | 32 | 30 | 25
hours | 0.525 [0.333 to 1.37] | 0.5 [0.417 to 1.42] | 0.5 [0.333 to 0.917]

4. Primary Outcome: Pharmacokinetic Analysis: Time to Maximum Concentration (Tmax) for Tolbutamide
Description: as for outcome 2
Time Frame: Baseline to 15 days post treatment
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Evaluable population.
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1: Tolbutamide Only | Part 1: Pexidartinib + Tolbutamide (Cycle 1, Day 1) | Part 1: Pexidartinib + Tolbutamide (Cycle 1, Day 11)
Number analyzed (Participants) | 32 | 30 | 25
hours | 2.90 [1 to 8.2] | 2.94 [1.52 to 8.08] | 3.17 [2.45 to 6.02]

5. Primary Outcome: Pharmacokinetic Analysis: Area Under the Curve to the Last Observable Concentration (AUClast) for Midazolam
Description: as for outcome 1
Time Frame: Baseline to 15 days post treatment
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Evaluable population.
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | Part 1: Midazolam Only | Part 1: Pexidartinib + Midazolam (Cycle 1, Day 1) | Part 1: Pexidartinib + Midazolam (Cycle 1, Day 11)
Number analyzed (Participants) | 32 | 30 | 25
ng*hour/mL | 43.7 (34.1) | 31.6 (19.6) | 18.5 (8.2)

6. Primary Outcome: Pharmacokinetic Analysis: Area Under the Curve to the Last Observable Concentration (AUClast) for Tolbutamide
Description: as for outcome 2
Time Frame: Baseline to 15 days post treatment
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Evaluable population.
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | Part 1: Tolbutamide Only | Part 1: Pexidartinib + Tolbutamide (Cycle 1, Day 1) | Part 1: Pexidartinib + Tolbutamide (Cycle 1, Day 11)
Number analyzed (Participants) | 32 | 30 | 25
ng*hour/mL | 500000 (196000) | 585000 (234000) | 700000 (207000)

7. Primary Outcome: Overall Summary of Treatment-emergent Adverse Events
Description: Adverse events that emerge during treatment, having been absent pre-treatment, or worsens relative to the pre-treatment state.
Time Frame: Baseline to 1 year post treatment
Population: Treatment-emergent adverse events (TEAEs) were assessed in the Safety Analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Drug-drug Interaction Phase | Part 2: Pexidartinib Only
Number analyzed (Participants) | 30 | 25
Participants
  TEAEs | 24 | 23
  Pexidartinib-related TEAEs | 16 | 20
  Treatment-emergent serious adverse events (SAEs) | 5 | 5
  Pexidartinib-related SAEs | 1 | 1

8. Secondary Outcome: Pharmacokinetic Analysis: Maximum Concentration (Cmax) for Pexidartinib and ZAAD-1006a Metabolite
Description: Plasma samples for pexidartinib and its metabolite were collected at predose, 0.5, 1, 2, 2.5, 3, 4, 6, 8, and 10 (±1) h after the first dose on Day 3, and at steady state when co-administered with midazolam and tolbutamide on Day 13.
Time Frame: Baseline to 13 days post treatment
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Evaluable population.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Part 1: Pexidartinib (Cycle 1, Day 1); Part 1: Pexidartinib (Cycle 1, Day 11): Pexidartinib was administered orally as a total daily dose of 800 mg (400 mg BID) starting from Day 3.
Arm/Group | Part 1: Pexidartinib (Cycle 1, Day 1) | Part 1: Pexidartinib (Cycle 1, Day 11)
Number analyzed (Participants) | 30 | 25
ng/mL
  Pexidartinib | 3140 (1250) | 8320 (2530)
  ZAAD-1006a | 3330 (1520) | 13500 (5980)

9. Secondary Outcome: Pharmacokinetic Analysis: Time to Maximum Concentration (Tmax) for Pexidartinib and ZAAD-1006a Metabolite
Description: as for outcome 8
Time Frame: Baseline to 13 days post treatment
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Evaluable population.
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1: Pexidartinib (Cycle 1, Day 1) | Part 1: Pexidartinib (Cycle 1, Day 11)
Number analyzed (Participants) | 30 | 25
hours
  Pexidartinib | 2.03 [1.08 to 7.83] | 1.93 [0.92 to 8.03]
  ZAAD-1006a | 6.04 [2.37 to 9.07] | 2.53 [0 to 8.25]

10. Secondary Outcome: Pharmacokinetic Analysis: Area Under the Curve to the Last Observable Concentration (AUClast) for Pexidartinib and ZAAD-1006a Metabolite
Description: as for outcome 8
Time Frame: Baseline to 13 days post treatment
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Evaluable population.
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | Part 1: Pexidartinib (Cycle 1, Day 1) | Part 1: Pexidartinib (Cycle 1, Day 11)
Number analyzed (Participants) | 30 | 25
ng*hour/mL
  Pexidartinib | 14400 (5870) | 53200 (17800)
  ZAAD-1006a | 18300 (7240) | 102000 (44100)

11. Secondary Outcome: Pharmacokinetic Analysis: Maximum Concentration (Cmax) for Midazolam Metabolite, 1-Hydroxy Midazolam
Description: Plasma samples for midazolam and 1-hydroxy midazolam were to be collected at predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8 (±10 min up to 8 h), 10 (±2), 24 (±2), and 48 (±2) hours on Days 1 to 3 and also when co-administered with pexidartinib on Days 3 to 5 and Days 13 to 15.
Time Frame: Baseline to 13 days post treatment
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Evaluable population.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1: Midazolam Only | Part 1: Pexidartinib + Midazolam (Cycle 1, Day 1) | Part 1: Pexidartinib + Midazolam (Cycle 1, Day 11)
Number analyzed (Participants) | 32 | 30 | 25
ng/mL | 49.7 (17.9) | 52.1 (17.4) | 55.7 (17.4)

12. Secondary Outcome: Pharmacokinetic Analysis: Time to Maximum Concentration (Tmax) for Midazolam Metabolite, 1-Hydroxy Midazolam
Description: as for outcome 11
Time Frame: Baseline to 13 days post treatment
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Evaluable population.
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1: Midazolam Only | Part 1: Pexidartinib + Midazolam (Cycle 1, Day 1) | Part 1: Pexidartinib + Midazolam (Cycle 1, Day 11)
Number analyzed (Participants) | 32 | 30 | 25
hours | 1.0 [0.333 to 1.45] | 0.933 [0.417 to 1.37] | 0.833 [0.383 to 1.55]

13. Secondary Outcome: Pharmacokinetic Analysis: Area Under the Curve to the Last Observable Concentration (AUClast) for Midazolam Metabolite, 1-Hydroxy Midazolam
Description: as for outcome 11
Time Frame: Baseline to 13 days post treatment
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Evaluable population.
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | Part 1: Midazolam Only | Part 1: Pexidartinib + Midazolam (Cycle 1, Day 1) | Part 1: Pexidartinib + Midazolam (Cycle 1, Day 11)
Number analyzed (Participants) | 32 | 30 | 25
ng*hour/mL | 200 (93) | 206 (95.5) | 212 (99.6)

14. Secondary Outcome: Pharmacokinetic Analysis: Metabolite to Parent Ratio (MPR) for Midazolam
Description: Plasma samples for midazolam were collected at predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 24, and 48 hours (h) (±10 minutes up to 1 h, ±10% thereafter) on Days 1 to 3, and also when co-administered with pexidartinib on Days 3 (to 5) and Days 13 (to 15).
  Plasma pharmacokinetic parameters calculated for Midazolam metabolite. 1-hydroxy midazolam and midazolam for the MPR value.
Time Frame: Baseline to 13 days post treatment
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Evaluable population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1: Midazolam Only | Part 1: Pexidartinib + Midazolam (Cycle 1, Day 1) | Part 1: Pexidartinib + Midazolam (Cycle 1, Day 11)
Number analyzed (Participants) | 32 | 30 | 25
Ratio | 587 (359) | 750 (391) | 1220 (657)

ADVERSE EVENTS:
Time Frame: Adverse events were collected after first dose up to 28 days after the last dose of study drug, up to 1 year.
Description: A treatment emergent adverse event (TEAE) was defined as an adverse event that emerges during treatment of Pexidartinib, having been absent pretreatment (Pexidartinib), or worsens relative to the pre-treatment (Pexidartinib) state.
Arm/Group | Part 1: Drug-drug Interaction Phase | Part 2: Pexidartinib Only
All-Cause Mortality (participants affected / at risk) | 1/30 | 0/25
Serious Adverse Events (participants affected / at risk) | 5/30 | 5/25
Other Adverse Events (participants affected / at risk) | 24/30 | 23/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Drug-drug Interaction Phase (N=30) | Part 2: Pexidartinib Only (N=25)
Pericardial effusion (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 1
Malignant bowel obstruction (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Pneumonia (Immune system disorders) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Drug-drug Interaction Phase (N=30) | Part 2: Pexidartinib Only (N=25)
Anemia (Blood and lymphatic system disorders) | 5 | 4
Eye swelling (Eye disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 3 | 3
Diarrhea (Gastrointestinal disorders) | 4 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 2 | 4
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 3
Chills (General disorders) | 2 | 1
Fatigue (General disorders) | 4 | 7
Alanine aminotransferase increased (Investigations) | 3 | 2
White blood cell count decreased (Investigations) | 1 | 6
Neutrophil count decreased (Investigations) | 0 | 4
Gamma-glutamyltransferase increased (Investigations) | 2 | 1
Blood lactate dehydrogenase increased (Investigations) | 2 | 0
Blood cholesterol increased (Investigations) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 5 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 4
Decreased appetite (Metabolism and nutrition disorders) | 2 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Headache (Nervous system disorders) | 2 | 1
Dysgeusia (Nervous system disorders) | 3 | 3
Dizziness (Nervous system disorders) | 1 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-28): https://cdn.clinicaltrials.gov/large-docs/88/NCT03291288/Prot_SAP_000.pdf